CLINICAL TRIAL: NCT02019186
Title: Effects of Vitamin C and E on Endothelial Function in Adolescent Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Robert Hoffman, Professor, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCRI-VITCE
Record Dates: First submitted 2013-12-18; First posted 2013-12-24 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes; endothelial function; adolescents; vitamin C; vitamin E
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Ascorbic Acid; Vitamin E

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vitamin C and E (Experimental): 6 weeks of daily treatment with Vitamin C and E
  Interventions: Dietary Supplement: Vitamin C; Dietary Supplement: Vitamin E

INTERVENTIONS:
Dietary Supplement: Vitamin C — <30 kg 250 mg 30-60 kg 500 mg >60 kg 750 mg
Dietary Supplement: Vitamin E — <30 kg 100 IU, 30-60 kg 200 IU, >60 kg 300 IU

SUMMARY:
The endothelium is the lining of the blood vessels that helps prevent damage to the vessels. The endothelium does not function as well as it should in adolescents with type 1 diabetes. This causes future diabetes complications. Adolescents with diabetes also have abnormalities of the cells that repair the endothelium. These abnormalities may be due to damage caused by intermittent hyperglycemia. This studied is designed to study whether low dose, combined Vitamin C and E supplementation improves endothelial function and repair in adolescents with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescent with T1D between 8 and 15 years of age will be studied.
2. Started on insulin therapy immediately after diagnosis.
3. Fasting c-peptide levels must be less than 0.4 ng/ml.
4. Hgb A1c levels greater than 8.3%.
5. All subjects must be in good health other than having diabetes. Subjects with hypothyroidism will be allowed assuming they are on stable thyroxine replacement and have normal thyroid function tests.
6. Females on oral contraceptives will also be eligible to participate.

Exclusion Criteria:

1. History oral hypoglycemic agent use.
2. BMI>95th percentile
3. Hypertension
4. Elevated creatinine levels
5. Microalbuminuria.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2013-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
endothelial function | 6 weeks
  Endothelial function will be measured before and after 6 weeks of therapy with Vitamin C and E

SECONDARY OUTCOMES:
Endothelial progenitor cells | 6 weeks
  Endothelial progenitor cells will be measured before and after 6 weeks of Vitamin C and E therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute at Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Hoffman RP, Dye AS, Bauer JA. Ascorbic acid blocks hyperglycemic impairment of endothelial function in adolescents with type 1 diabetes. Pediatr Diabetes. 2012 Dec;13(8):607-10. doi: 10.1111/j.1399-5448.2012.00882.x. Epub 2012 Aug 28. PMID 22925199
- [Background] Dye AS, Huang H, Bauer JA, Hoffman RP. Hyperglycemia increases muscle blood flow and alters endothelial function in adolescents with type 1 diabetes. Exp Diabetes Res. 2012;2012:170380. doi: 10.1155/2012/170380. Epub 2012 Jun 3. PMID 22701470
- [Background] Varvarovska J, Racek J, Stozicky F, Soucek J, Trefil L, Pomahacova R. Parameters of oxidative stress in children with Type 1 diabetes mellitus and their relatives. J Diabetes Complications. 2003 Jan-Feb;17(1):7-10. doi: 10.1016/s1056-8727(01)00228-8. PMID 12505749